CLINICAL TRIAL: NCT02345421
Title: A Study to Identify the Frequency of Lysosomal Acid Lipase Deficiency in At-Risk Patient Populations
Brief Title: A Study to Identify and Characterize LAL-D Patients in High-risk Populations
Status: Terminated | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LAL-CSS01
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Lysosomal Acid Lipase Deficiency
Keywords: LAL D; CESD; NASH; NAFLD; Wilson's; Niemann Pick; Familial Hypercholesterolemia
MeSH Terms: conditions — Wolman Disease; Non-alcoholic Fatty Liver Disease; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- At risk population

SUMMARY:
The objective of this study is to determine the frequency of Lysosomal Acid Lipase Deficiency (LAL D) by lysosomal acid lipase (LAL) enzyme activity assay in patients who are considered to be at risk.

ELIGIBILITY:
Inclusion Criteria:

1. Non-obese** patients with elevated low-density lipoprotein (LDL)
2. Non-obese** patients with low high-density lipoprotein (HDL)
3. Non-obese** patients with unexplained and persistently elevated liver transaminases,
4. Non-obese** patients with hepatomegaly
5. Patients with cryptogenic cirrhosis
6. Patients with biopsy-proven microvesicular or mixed micro/macrovesicular steatosis without a known etiology
7. Patients with presumed Familial Hypercholesterolemia (FH) in which genetic analysis was performed for the genes encoding the low-density lipoprotein receptor (LDLR), Apo-B and PCSK9 genes and no disease-causing mutations were identified
8. Patients with presumed FH with unclear family history
9. Patients with autosomal recessive hypercholesterolemia (other than homozygous FH)
10. Patients with autosomal recessive low HDL of unknown etiology

Also, patient must meet the following:

* Patient or patient's parent or legal guardian (if applicable) consents to participate in the study and provides informed consent prior to any study procedures being performed. If the patient is of minor age; he/she is willing to provide assent where required per local regulations, and if deemed able to do so.
* Patient is willing and able to comply with protocol requirements.
* Patients who do not fall into one of the aforementioned categories (cohorts) but are considered highly suspicious for LAL D should be tested to rule out the disorder outside of the study at the discretion of the Investigator.

Exclusion Criteria:

* Active viral hepatitis;
* Other confirmed genetic liver diseases (e.g., Wilson's disease, hemochromatosis, alpha 1-antitrypsin).

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients >2 years of age who are at risk for a diagnosis of LAL D
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
LAL D frequency based on LAL enzyme assay. | approximately 1 month
  The endpoint of this study is the frequency of LAL D in at-risk patients, based on results from the LAL enzyme assay.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - San Francisco, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Orleans, Louisiana
  - Minneapolis, Minnesota
  - The Bronx, New York
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Houston, Texas
  - San Antonio, Texas